CLINICAL TRIAL: NCT03331523
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Calcipotriene and Betamethasone Dipropionate Topical Suspension, 0.005%/0.064% (Glenmark Pharmaceuticals Ltd) to the Marketed Product Taclonex® Topical Suspension (LEO Pharma Inc.) in the Treatment of Scalp Psoriasis
Brief Title: To Study Generic Calcipotriene and Betamethasone Dipropionate Topical Suspension, 0.005%/0.064%, in the Treatment of Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLK-1701
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Scalp Psoriasis
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Calcipotriene/betamethasone dipropionate (Experimental)
  Interventions: Drug: Calcipotriene/Betamethasone Dipropionate
- Taclonex® (Active Comparator)
  Interventions: Drug: Taclonex®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcipotriene/Betamethasone Dipropionate — Topical suspension 0.005%/0.064% (Glenmark Pharmaceuticals Ltd)
  Arms: Calcipotriene/betamethasone dipropionate
Drug: Taclonex® — Calcipotriene/ betamethasone dipropionate topical suspension, 0.005%/0.064% (LEO Pharma Inc.)
  Arms: Taclonex®
Drug: Placebo — Placebo of Calcipotriene/ betamethasone dipropionate topical suspension, 0.005%/0.064% (Glenmark Pharmaceuticals Ltd.)
  Arms: Placebo

SUMMARY:
This is a phase III, randomized, double-blind, placebo-controlled, parallel- group, multiple-site study to evaluate the therapeutic equivalence of generic calcipotriene and betamethasone dipropionate topical suspension, 0.005%/0.064% of Glenmark Pharmaceuticals Ltd to that of the marketed product Taclonex® topical suspension of Leo Pharma Inc. in the treatment of scalp psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female subjects aged at least 18 years at Visit 1.
2. A clinical diagnosis of stable (at least 6 months) scalp psoriasis involving at least 10% of the scalp and clinical signs of psoriasis vulgaris on trunk and/or limbs.
3. A PGA of disease severity of the scalp psoriasis consistent with at least moderate disease severity (Grade ≥ 3).
4. A plaque elevation of at least moderate severity (Grade ≥ 3) at the scalp target lesion site. The most severe scalp lesion at baseline should be identified as the target lesion.

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative, or pustular psoriasis.
2. Other inflammatory skin disease in the scalp that may confound the evaluation of the scalp psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea capitis).
3. Presence of pigmentation, extensive scarring, pigmented lesions, or sunburn in the scalp that could interfere with the rating of efficacy parameters.
4. Presence of viral lesions, fungal, bacterial, or parasitic infections and/or atrophic (thinning) skin on the scalp.
5. History of psoriasis unresponsive to topical treatments.
6. Subjects with planned phototherapy and/or exposure to ultraviolet A (UVA) and/or UVB during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each treatment group with treatment success, defined as a score of 0 or 1, within the treatment area(s) on the PGA scale of disease severity, at the end of study visit. | Day 29
Proportion of subjects in each treatment group with clinical success, defined as a score of 0 or 1, at the target lesion site on the PASI scale at the end of study visit. | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: William Todd Kays, Study Director — Glenmark Pharmaceuticals Inc., USA
Locations (31):
- United States (31):
  - Investigational Site 24, Encinitas, California
  - Investigational Site 3, Fremont, California
  - Investigational Site 13, San Diego, California
  - Investigational Site 20, San Diego, California
  - Investigational Site 32, Santa Monica, California
  - Investigational Site 14, Denver, Colorado
  - Investigational Site 1, Miami, Florida
  - Investigational Site 30, Miami, Florida
  - Investigational Site 7, Miramar, Florida
  - Investigational Site 22, Tampa, Florida
  - Investigational Site 15, New Albany, Indiana
  - Investigational Site 10, South Bend, Indiana
  - Investigational Site 21, Louisville, Kentucky
  - Investigational Site 6, Ann Arbor, Michigan
  - Investigational Site 12, Fridley, Minnesota
  - Investigational Site 26, Saint Joseph, Missouri
  - Investigational Site 17, Henderson, Nevada
  - Investigational Site 25, Las Vegas, Nevada
  - Investigational Site 29, Forest Hills, New York
  - Investigational Site 28, Rochester, New York
  - Investigational Site 4, High Point, North Carolina
  - Investigational Site 18, Fountain Inn, South Carolina
  - Investigational Site 27, Mt. Pleasant, South Carolina
  - Investigational Site 9, Knoxville, Tennessee
  - Investigational Site 8, Nashville, Tennessee
  - Investigational Site 5, Austin, Texas
  - Investigational Site 11, College Station, Texas
  - Investigational Site 16, San Antonio, Texas
  - Investigational Site 19, San Antonio, Texas
  - Investigational Site 31, Norfolk, Virginia
  - Investigational Site 23, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No